CLINICAL TRIAL: NCT05426226
Title: Effect of Low Level Light Irradiation on Insomniacs' Meridians During the First Sleep Cycle.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, vghtpe user, Center for Traditional Medicine,Attending Doctor, Principal Investigator,, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB 2022-02-027B
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Insomnia
Keywords: Heart rate variability; meridian; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The subjects were randomly assigned to group A and group B, the group A will take light acupuncture in the first month, and sham in the next month; Group B is opposite.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants allocation by third party
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser group (Active Comparator): Laser group use specific wavelength to light the sleep acupoints during.
  If the laser group take light acupuncture in the first month, and then become the sham group in the next month, vice versa.
  Interventions: Device: laser acupuncture
- sham group (Sham Comparator): sham group use the same divce and acupointsas the laser group, but the light is just a regular light.
  If the laser group take light acupuncture in the first month, and then become the sham group in the next month, vice versa.
  Interventions: Device: sham device

INTERVENTIONS:
Device: laser acupuncture — using laser acupuncture device on sleep acupoints during sleep
  Arms: laser group
Device: sham device — using sham device on sleep acupoints during sleep
  Arms: sham group

SUMMARY:
Introduction In the past, it was found that stimulating the meridians and acupoints with low-level light often had a good effect. However, for safety reasons, most instruments such as laser acupuncture devices still need to be used by medical personnel, and it is difficult to apply to insomnia patients at bed-time or the first sleep cycle, these two periods have a considerable impact on sleep quality.

Therefore, the purpose of this study is to provide a safer wearable light-therapy device for Insomnia patients, so that it can be used in home sleep situations, and the improvement of subjects' sleep qualtity and meridian energy will be evaluated by PSG, HRV parameters, sleep questionnaires, and Ryodoraku value (reflects the meridian electric resistance).

Methods Aim1: To evaluate whether the subjects are more relaxed by observing the changes in heart rate and meridian energy of healthy subjects after low-level light irradiating to Shenmen, Daling, Neiguan (acupoints for insomnia). We also consider the difference of light source and the skin color in experiment design. Aim2: To assess whether the insomnia patients' sleep quality has improved after applying the wearable light therapy device to subjects' bed-time (include the first sleep cycle). We use PSG, sleep questionnaires, stroop test for evaluation.

DETAILED DESCRIPTION:
Hypotheses and Aims

In the past, there are no studies on using light acupuncture during the first sleep cycle or bed-time. So, we have the following hypotheses: First, irradiating low level light on the sleep acupoints during these periods will strengthen the activity of the parasympathetic during these periods; Second, the activity of the parasympathetic will improve the quality of sleep in the first sleep cycle, because the parasympathetic activity of sleep onset(SO) is an indicator of sleep quality; Third, the improvement of sleep quality in the first sleep cycle will affect the quality of total sleep and daytime cognitive functions. I divide the research hypotheses for details into three categories:

Part 1: To observe the relationship between light stimulation of traditional Chinese medicine (TCM) sleep-aiding acupoints.

Hypothesis 1-1: After the laser stimulates the sleep-aiding acupoints, the energy of the meridian that is too high will decrease, and the energy of the meridian that is too low will increase.

Hypothesis 1-2: After laser acupuncture, the qi of the meridians will not be consumed too quickly like acupuncture, so the needle retention is safe.

Hypothesis 1-3: The efficacy of LED stimulation of acupoints should be similar to that of laser acupuncture.

Part 2: Assumptions Related to Optical Design:

Hypothesis 2-1: The most suitable light specifications for dark-skinned people are different from light-skinned people.

Hypothesis 2-2: Some new optical components have good performance in light transmission Hypothesis 2-3: The newly designed light penetration experiment can obtain optical parameters more accurately and quickly

Part 3: Heart Rate Variability and Sleep Improvement:

Hypothesis 3-1: We could improve parameters of heart rate variability by using the wearable light therapy device.

Hypothesis 3-2: Optimizing HRV parameters before going to bed can improve the quality of the first sleep cycle.

Hypothesis 3-3: After using a wearable light therapy device to improve the first sleep cycle, it can also enhance the whole night sleep quality.

Hypothesis 3-4: Improved sleep quality from using wearable light therapy device can lead to the improvements in daily cognitive function.

Significance If this study is successfully proved to improve the sleep quality of insomnia patients, it will give insomnia patients a treatment option other than sleep pills, make light therapy be widely applied to the home environment, and make researchers pay more attention to the possibility of using TCM procedure in the first sleep cycle.

Research Materials and Equipment Research Methods

STAGE 1:

Participant

Experiment A:

A preliminary experiment of "laser acupuncture" on sleep acupoints (healthy subjects).

Subjects: 30 healthy subjects.

Designs

Experimental procedure:

1. The experiments will be carried out twice, once with laser intervention, and once with sham. The experiment time was 25 minutes, and both were scheduled between 3:30 and 5:00 PM. The room temperature was controlled between 25-27 degrees. The interval between two experiments is between one to two weeks to avoid the influence of seasonal factors.
2. Before the experiment, the subjects' Ryodoraku value will be measured. The subjects shall sit in a fixed posture and step on the square box at room temperature and avoid touching metal or cold materials.
3. Before the start of the experiment, ask the subject to hold the hand-held heart rate measurement device and teach him how to use it; set up the laser acupuncture head on the sleep acupoints we used; then blindfold him with a blinder.
4. From 0 to 5 minutes, let the subject measure the first HRV parameters as the data [before intervention].
5. From the 5th to 10th minute of the experiment, the laser or sham intervenes at the eighth minute, and the intervention time lasts for ten minutes.
6. From the 10th to 15th minute, the subject measured the second time HRV parameters, which was used as the data of the [during the intervention].
7. In the 15th to 20th minutes, the laser or sham will end the intervention at the 17th to 18th minutes.
8. From the 20th to 25th minute of the experiment, the subject measured the third heart rate variability parameters under blindfolded conditions, as the data of the [after the intervention].
9. Take off his blinder, Ask the subject to measure Ryodoraku value again, and end the experiment.

   * Sham intervention method: The subject in blindfolded state can hear the same prompt sound as laser acupuncture, but does not irradiate light. (Fig.3-4)

Experiment B: All procedures are the same as Experiment A, but the light source is change to LED wearable devices. (Fig.5-6)

STAGE 2:

Participant Subjects: 120 insomnia subjects. (80 subjective insomnia; 40 objective insomnia)

Designs

Experimental procedure:

Prepare period:

1. Inform the subjects of the research process, complete questionnaire such as PSQI, MEQ, ISI, ESS, and limb motor sensory survey to determine whether they are eligible for the study.
2. The subject fills in the sleep diary for one week and wears an oximeter to confirm that there is no sleep abnormality.
3. The subject used a tiny wireless sleep physiological recorder to record the quality of sleep for two nights. The first night was the adaptation period and was not included in the analysis, and the sleep data of the second night was included in the analysis (base line).

Experimental period:

1. DAY0: The subjects were randomly assigned to group A and group B, the group A will take light acupuncture in the first month, and sham in the next month; Group B is opposite.
2. DAY1: The subject filled out the rest of the questionnaires, and then asked them to complete the Ryodoraku measurement, and wear the TD1 tiny PSG recorder to perform the first multi-channel physiological measurement, explain the use process of the wearable light therapy deivce, and let them download the EncephalApp stroop test Program.
3. DAY15: All procedures are the same as DAY1, but no questionnaires. (second tiny PSG record)
4. DAY30: All procedures are the same as DAY1, fill questionnaires like PSQI, ISI etc. (third tiny PSG record)
5. DAY31-DAY36: take a break and do nothing.(wash-out)
6. DAY37: All procedures are the same as DAY1. (fourth tiny PSG record)
7. DAY52: All procedures are the same as DAY15. (fifth tiny PSG record)
8. DAY67: All procedures are the same as DAY30. (sixth tiny PSG record)
9. DAY68: The subject returned the wearable light therapy device and TD1 recorder, and confirmed whether the data of TD1 is complete. (Fig. 7)

Analysis Methods The main data is expressed in terms of mean and standard deviation (SD). The before -after difference in same groups is analyzed by t-test, and the difference between groups is also analyzed by ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 to 65 years
* No sleep pills for 3 months
* Body Mass Index (BMI) : 18.5-30
* Blood pressure: within normal range (140 mmHg/90 mmHg)
* People with regular wake-up time
* The bedtime is between 22:00 and 2:00.

Exclusion Criteria:

* People with sleep disorders other than insomnia
* those currently taking drugs;
* with cardiovascular disease, cancer, psychiatric disease, kidney disease, diabetes, chronic disease and physical discomfort
* Exclude tobacco, alcohol, caffeine, and drug addicts
* Exclude from fitzpatrick skin type classification - V and VI (skin is black and dark brown)
* People whose skin is allergic to light (light sensitivity, solar dermatitis).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-10 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Differences in sleep EEG before and after the laser irradiation compared to the sham group | Change from Baseline sleep EEG at 67 days
  According to sleep EEG,we can analysis participants' brain waves (alpha,beta,theta,delta) and sleep stages,etc. to evaluate their objective sleep quality
Differences in Heart rate variability before and after the laser irradiation compared to the sham group | Change from heart rate variability parameters at 67 days
  HRV is measured by the variations in the R-R interval between the successive peaks of the QRS complex in the ECG wave. Based on fast Fourier transform, time-domain (R-R interval) transfer to frequency domain resulting total power (TP, 0.04-0.15), low frequency (LF, 0.06-0.6Hz), high frequency (HF, 0.6-2.4Hz), normalized LF (LF%) and LF/HF ratio are obtained. LF% and HF represent an index of sympathetic activity and parasympathetic activity respectively. LF/HF is indicative of the sympathetic to parasympathetic autonomic balance.

SECONDARY OUTCOMES:
Differences in the Epworth Sleepiness Scale (ESS) before and after the laser irradiation compared to the sham group. | Change from Baseline ESS at 67 days
  The Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subje
Differences in Visual Analogue Scale (VAS) before and after the laser irradiation compared to the sham group. | Change from Baseline VAS at 67 days
  Visual Analogue Scale (VAS) consists of a line, 10 cm in length. Individuals point to or mark a spot on the line where they feel indicates their current their emotion, fatigue level and sleep quality. The score of emotion level is from 0cm (very nervous) to 10 cm (very relaxing). The score of fatigue level is from 0 cm (very energetic) to 10 cm (very sleepy). The score of sleep quality is from 0 cm (poor) to 10 cm (sleep well). The maximum total score is 100% (equal 10cm).
Differences in scores of stroop test before and after the laser irradiation compared to the sham group. | Change from Baseline score of stroop at 67 days
  The Visual Stroop Test is designed to assess cognitive flexibility and attention span by examining a patient's ability to separate word and color naming stimuli through the use of three separate subtests.
Differences in the Insomnia Severity Index (ISI) before and after the laser irradiation compared to the sham group. | Change from Baseline ISI at 67 days
  Designed as a brief screening tool for insomnia, the seven-item questionnaire asks respondents to rate the nature and symptoms of their sleep problems using a Likert-type scale. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia.The maximum total score is 28.
Differences in the Pittsburgh sleep quality index before and after the laser irradiation compared to the sham group. | Change from Baseline PSQI at 67 days
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.The maximum total score is 21. A higher score reflects more poor sleep quality.
Differences in The Beck Depression Inventory II (BDI-II) before and after the laser irradiation compared to the sham group. | Change from Baseline BDI-II at 67 days
  The Beck Depression Inventory II (BDI-II) is a 21-item, self-rated scale that evaluates key symptoms of depression. It rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. A higher score reflects greater symptoms of depression.
Differences in Beck Anxiety Inventory (BAI) before and after the laser irradiation compared to the sham group. | Change from Baseline BAI at 67 days
  the Beck Anxiety Inventory (BAI) is a 21-item, self-rated scale that evaluates anxiety levels , rated on a scale from 0 to 3. Each item is descriptive of subjective, somatic, or panic-related symptoms of anxiety.The maximum total score is 63.A higher score reflects greater anxiety.
Differences in Chinese 14-item PSS before and after the laser irradiation compared to the sham group. | Change from Baseline PSS at 67 days
  The PSS is an 14-item instrument designed to measure the perception of stress in a month . All items are rated on a 5-point Likert scale from 0 (never) to 4 (very often) and seven of them (4, 5, 6, 7, 9, 10, 13) are reverse-scored.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Pu Tseng, MD, Principal Investigator — Center for Traditional Medicine
Locations (1):
- Center for Traditional Medicine, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No